CLINICAL TRIAL: NCT04322630
Title: Detecting Soluble MER Levels After Myocardial Ischemia and Reperfusion Injury in Pediatric Patients
Brief Title: Mer-TK in Human Cardiac Cells
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-2445
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Myocardial Inflammation; Myocardial Infarction
MeSH Terms: conditions — Myocarditis; Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Human blood samples obtained intra-operatively during cardiac bypass.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Cardiac Bypass Patients: Blood samples obtained from patients ages from birth-19 years-old as well as cyanotic and acyanotic cardiac lesions who underwent cardiac bypass.
  Interventions: Other: Change in Soluble MER Concentration

INTERVENTIONS:
Other: Change in Soluble MER Concentration — Measuring change in soluble MER Concentration post compared to pre bypass for each patient.

SUMMARY:
The relationship between the immune system and the myocardium after myocardial ischemia is an evolving field of research. Crosstalk occurs between macrophages and cardiac myocytes to promote cardio-protection and resolution of inflammation after myocardial ischemia and reperfusion injury (MI/R injury).

Myeloid-epithelial-reproductive tyrosine kinase (MerTK), a member of the TAM family of tyrosine kinase receptors (Tyro-Axl-MerTK), is a macrophage receptor that mediates efferocytosis, anti-inflammatory signaling, and resolution of inflammation. After MI/R injury, intact MerTK is necessary for the phagocytosis of dead cardiac myocytes and to promote anti-inflammatory signaling. Proteolytic cleavage of MerTK to its inactive form, soluble MER, restricts the capacity of macrophages to phagocytize dead cardiac myocytes and impairs MerTK-dependent anti-inflammatory signaling resulting in suppressive effects on cardiac remodeling and function.

The Thorp lab at Northwestern University has previously measured soluble MER levels in both adult mice and humans and found that soluble MER concentrations increase after MI/R injury. In adult MI patients, soluble MER was measured post coronary artery reperfusion and was found to be increased (average 3200 pg/mL compared to 1700 pg/mL) compared to controls with stable cardiovascular disease. Based on murine data, the lab further postulated that reperfusion injury may directly interfere with MerTK-dependent cardiac repair as reactive oxygen species formed during reperfusion injury induce proteolytic cleavage of MerTK to soluble MER.

Myocardial infarctions are rare events in pediatric patients. However, pediatric hearts are exposed to periods of hypoperfusion, ischemia, and inflammation during times of stress such as cardiac bypass and critical illness, and it is unknown how soluble MER levels change in response to these events. Thus, I was interested in investigating how soluble MER levels change after MI/R injury induced by cardiac bypass as well as in the utility of soluble MER as a biomarker of cardiac inflammation and injury in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* All patient ages from birth-19 years-old as well as cyanotic and acyanotic cardiac lesions will be included

Exclusion Criteria:

* Patients will be excluded if both pre and post bypass blood samples are not available.

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with congenital heart disease presenting to Lurie Children's Hospital for corrective or palliative heart surgery and will be undergoing cardiac bypass.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Soluble MER Concentration | 5/10/2019-12/31/2020

SECONDARY OUTCOMES:
Utility of soluble MER as a biomarker of inflammation and injury | 5/10/2019-12/31/2020

CONTACTS AND LOCATIONS:
Locations (1):
- Ann & Robert H Lurie Children's Hopsital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided